CLINICAL TRIAL: NCT02898389
Title: Influence of Chronic Vascular Diseases on Transcranial Doppler Profiles in Critically Ill Patients
Acronym: CritiDop
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/LM-01b; NCT03043092 (obsolete NCT alias)
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Respiration, Artificial; Sedated
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: With cardiovascular risk factors: Patients fall within this group when they have at least one of the cardiovascular risk factors listed in the eligibility criteria section.
- Group 1: Without cardiovascular risk factors: Patients fall into this group when they do not have any of the cardiovascular risk factors listed in the eligibility criteria section.

SUMMARY:
The primary objective of this study is to show that cardiovascular risk factors associated with the chronic elevation of arterial resistance may be associated with "false" profiles of intracranial hypertension during transcranial doppler ultrasound of the middle cerebral arteries in intensive care unit patients. A "false" profile of intracranial hypertension is defined by a high pulsatility index without any intracranial pathology.

ELIGIBILITY:
Inclusion Criteria for entry in the study:

* Sedated patient under mechanical respiratory assistance

Inclusion criteria for entry in group 1: the patient meets at least one of the following criteria:

* The patient is a man over the age of 50 or a woman over the age of 60
* Hypercholesterolemia (LDL > 1.6 g/L, HDL < 0.4 g/L)
* Arterial hypertension for over 10 years (treated or systolic arterial pressure > 140 mmHG)
* Type 2 diabetes for over 10 years
* Active or former smoker in the past 3 years
* History of cardiovascular event (peripheral artery disease, heart attack, stroke/transient ischemic attack over 3 months ago)
* Chronic renal insufficiency with MDRD < 30 ml/min/1.73m^2

Inclusion criteria for entry in group 2:

* The included patient is not in group 1

Exclusion Criteria:

* acute neurological disorder (brain trauma, infectious or immune meningitis, meningoencephalitis, ischemic or hemorrhagic stroke <3 months)
* pregnant woman
* person under guardianship
* prisoners
* recent carotid surgery (<1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sedated patients under mechanical respiratory assistance will be included. These are further devided into 2 groups.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Pulsatility index on the middle cerebral arteries | Day 0
Diastolic velocity at the middle cerebral arteries | Day 0
Mean velocity at the middle cerebral arteries | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Muller, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France